CLINICAL TRIAL: NCT00997243
Title: Phase II Study of 5-azacytidine and Lintuzumab in Myelodysplastic Syndromes (MDS)
Brief Title: Azacitidine and Lintuzumab in Treating Patients With Previously Untreated Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug no longer being supplied by sponsor
Sponsor: Alison Walker (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor-Investigator, Alison Walker, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-09034; NCI-2011-03159 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Results first posted 2013-11-26 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-04

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: de novo myelodysplastic syndromes; secondary myelodysplastic syndromes; chronic myelomonocytic leukemia; refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; refractory anemia with ringed sideroblasts; refractory anemia; refractory cytopenia with multilineage dysplasia
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Anemia, Refractory, with Excess of Blasts; Anemia, Refractory | interventions — lintuzumab; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 5-azacytidine and Lintuzumab (Experimental): Cycle 1- 5-azacytidine (Vidaza, AZA) 75mg/m2 IV/SC(subcutaneous)daily on days 1-7.
  Subsequent Cycles (cycles to be repeated every 28 days) AZA 75mg/m2 IV/SC daily on days 1-7.
  Interventions: Biological: lintuzumab; Drug: 5-azacytidine

INTERVENTIONS:
Biological: lintuzumab — Cycle 1 600mg as an IV infusion (flat dose for all), given on days 2, 7, 15, and 22. Subsequent Cycles (cycles to be repeated every 28 days) 600mg as an IV infusion, given every other week, twice during each cycle, including one dose given during AZA therapy. Doses should be given at least 12 days apart. By convention, dosing on days 7 and 22 of each cycle will be encouraged, but due to expected issues of patient convenience (time, travel, etc.), the study requirements are every other week, twice during each cycle, with one dose during AZA treatment.
  Other Names: SGN-33
Drug: 5-azacytidine — 75mg/m2 IV/SC daily on days 1-7.
  Other Names: Vidaza; AZA

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as lintuzumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving chemotherapy together with monoclonal antibodies may be a better way to block cancer growth.

PURPOSE: This phase II trial is studying the side effects and how well giving azacitidine together with lintuzumab works in treating patients with previously untreated myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the complete response rate of the combination of lintuzumab and azacitidine in patients with myelodysplastic syndromes.

Secondary

* To define the specific toxicities of this regimen.
* To determine the overall response rate.
* To determine the relationship between pretreatment expression of Syk and clinical response.
* To determine whether the investigational agents modulate Syk expression and to correlate drug-induced changes in Syk with response to treatment.
* To provide preliminary data on the biological activity of azacitidine as a demethylating agent (changes in target gene methylation and gene expression, DNMT1 protein expression, global methylation).
* To perform exploratory studies of azacitidine-triphosphate with global DNA methylation.
* To explore the biologic role of microRNA in determining clinical response to this regimen and achievement of the other pharmacodynamic endpoints.

OUTLINE: Patients receive azacitidine IV or subcutaneously once daily on days 1-7 and lintuzumab IV on days 2, 7, 15, and 22 (days 2 and 15 of course 1 only). Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. Treatment modifications may apply according to response.

Blood and bone marrow samples are collected periodically for pharmacodynamic studies.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Eligibility Criteria:

* Age >18 with untreated MDS by FAB or WHO criteria (note: FAB criteria for MDS includes <29% blasts; FAB criteria includes CMML).
* Patients with therapy related disease (t-MDS).
* If the patient has co-morbid medical illness, life expectancy attributed to this must be greater than 6 months.
* Eastern Cooperative Oncology Group (ECOG) performance status <2.
* Must have adequate organ function as defined below:

  * total bilirubin <2.0mg/dL
  * AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
  * creatinine <2.0mg/dL
  * NYHA CHF(congestive heart failure)Class II or better
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence).
* Ability to understand and willingness to sign the written informed consent document.
* CD33 expression is required on at least 25% of left shifted dysplastic myeloid cells, including blasts. This testing will be done on bone marrow aspirate, but for patients whose CD33 expression in this cellular compartment cannot be ascertained, peripheral blood will be allowed to determine this.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 6 months (for other cancers) prior to entering the study.
* Patients receiving any other investigational agents or patients that have received other investigational agents within 1 month of enrollment.
* Patients with active central nervous system disease or with granulocytic sarcoma as sole site of disease.
* Patients with history of allergic reactions attributed to compounds of similar chemical or biologic composition to AZA or lintuzumab that are not easily managed are excluded. Patients with hypersensitivity to mannitol are excluded.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. As infection is a common feature of MDS, patients with active infection are permitted to enroll provided that the infection is under control. Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Psychiatric conditions that prevent compliance with protocol or consent.
* Pregnant women or women who are breastfeeding are excluded from this study.
* HIV-positive patients on combination antiretroviral therapy are ineligible.
* Patients with serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Patients with serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Patients with baseline fibrinogen <100mg/dL, or those with clinically significant disseminated intravascular coagulation, are excluded.
* Patients who require ongoing therapeutic anticoagulation with warfarin, lovenox, or similar agent are excluded. This does not apply to patients on low dose prophylaxis therapy.
* Patients who require ongoing clopidogrel therapy are excluded. In cases where clopidogrel use at screening is subsequently discontinued due to ongoing or future risk of drug and treatment related cytopenias, such patients will be eligible.
* Patients with platelet <10,000/uL who are refractory to platelet transfusion are not eligible (must bump to at least >10,000/uL after transfusion)
* Patients who have previously received lenalidomide or thalidomide are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2010-09 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Walker, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- 5-azacytidine and Lintuzumab: Cycle 1- 5-azacytidine (Vidaza, AZA) 75mg/m2 IV/SC daily on days 1-7.
  Subsequent Cycles (cycles to be repeated every 28 days) AZA 75mg/m2 IV/SC daily on days 1-7.
Period: Overall Study
Arm/Group | 5-azacytidine and Lintuzumab
Started | 7
Completed | 0
Not Completed | 7
Not completed — Early termination of study by sponsor | 7

BASELINE CHARACTERISTICS:
Groups:
- 75 mg/m2 5-azacytidine (Vidaza, AZA) and 600 mg Lintuzumab: 5-azacytidine (Vidaza, AZA) 75mg/m2 IV/SC daily on days 1-7 cycle 1 and all subsequent cycles. Lintuzumab 600mg as an IV infusion (flat dose for all), given on days 2, 7, 15, and 22 for cycle 1 and 600mg as an IV infusion, given every other week, twice during each cycle, including one dose given during AZA therapy for all other subsequent cycles.
Arm/Group | 75 mg/m2 5-azacytidine (Vidaza, AZA) and 600 mg Lintuzumab
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: Response to therapy was determined based on percentage of blasts in bone marrow, hematopoiesis, and requirement for supportive care (i.e., transfusions or cytokine growth factors). The modified International Working Group response criteria was used, based on Cheson, et al.
Time Frame: up to 5 years
Measure: Number; unit: percentage of participants
Arm/Group | 5-azacytidine and Lintuzumab
Number analyzed (Participants) | 7
percentage of participants | 14

2. Secondary Outcome: Overall Response Rate
Description: as for outcome 1
Time Frame: up to 5 years
Measure: Number; unit: percentage of participants
Arm/Group | 5-azacytidine and Lintuzumab
Number analyzed (Participants) | 7
percentage of participants | 14

3. Secondary Outcome: Toxicities of the Combination
Description: All patients who received study drug were closely monitored for adverse events (AEs). All AEs that occured during study period were reported and the investigator determined the severity and relationship to study drug (unrelated, unlikely, possibly, probably, or definitely related). The NCI's CTCAE(Common Toxicity Criteria for Adverse Effects)v3.0 was used for grading AEs.
Time Frame: up to 5 years
Measure: Number; unit: percentage of participants
Arm/Group | 5-azacytidine and Lintuzumab
Number analyzed (Participants) | 7
percentage of participants
  Thrombosis/embolism (vascular access-related) | 14
  Platelets | 100
  Neutrophils/granulocytes (ANC/AGC) | 100
  Lymphopenia | 57
  Leukocytes (total WBC) | 100
  Infection with unknown ANC - Upper airway NOS | 14
  Infection with normal ANC or Grade 1 or 2 neutroph | 14
  Infection with unknown ANC - Bladder (urinary) | 14
  Infection | 28
  Infection Grade 3 or 4 neutrophils-blood | 28
  Hemorrhage, GI (lower GI NOS/Rectum) | 14
  Hemorrhage/Bleeding - Other | 14
  Hemoglobin | 100
  Fever (in the absence of neutropenia) | 28
  Febrile neutropenia (fever of unknown origin) | 14

4. Secondary Outcome: Determine the Relationship Between Pretreatment Expression of Syk and Clinical Response; to Determine Whether the Investigational Agents Modulate Syk Expression and Correlate Drug-induced Changes in Syk With Response to Treatment
Time Frame: up to 5 years
Population: No participants were analyzed due to withdrawal of the investigational agent by the company.
Arm/Group | 5-azacytidine and Lintuzumab
Number analyzed (Participants) | 0

5. Secondary Outcome: Provide Preliminary Data on the Biological Activity of AZA as a Demethylating Agent (Changes in Target Gene Methylation and Gene Expression, DNMT1[Deoxyribonucleic Acid Methyltransferase 1 DNA Methyltransferase 1]Protein Expression, Global Methylation)
Time Frame: up to 5 years
Population: No participants were analyzed due to withdrawal of the investigational agent by the company.
Arm/Group | 5-azacytidine and Lintuzumab
Number analyzed (Participants) | 0

6. Secondary Outcome: Perform Exploratory Studies of AZA-triphosphate With Global DNA Methylation
Time Frame: up to 5 years
Population: No participants were analyzed due to withdrawal of the investigational agent by the company.
Arm/Group | 5-azacytidine and Lintuzumab
Number analyzed (Participants) | 0

7. Secondary Outcome: Explore the Biologic Role of microRNAs in Determining Clinical Response to the AZA Plus Lintuzumab Combination and Achievement of the Other Pharmacodynamic Endpoints
Time Frame: Up to 5 years
Population: No participants were analyzed due to withdrawal of the investigational agent by the company.
Arm/Group | 5-azacytidine and Lintuzumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include events present at screening and after discontinuation from study (day 30).
Arm/Group | 5-azacytidine and Lintuzumab
Serious Adverse Events (participants affected / at risk) | 7/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-azacytidine and Lintuzumab (N=7)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cystitis (Hepatobiliary disorders) | 1 (1)
Distension/bloating, abdominal (Gastrointestinal disorders) | 2 (3)
Dizziness (Nervous system disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Edema: limb (General disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 (5)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Blood and lymphatic system disorders) | 1 (2)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2 (3)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage, GI - Lower GI NOS (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 1 (1)
Hemorrhage/Bleeding - Other (Specify, __) (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e (Infections and infestations) | 1 (1) — Blood
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e (Infections and infestations) | 1 (1) — Mucosa
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e (Infections and infestations) | 1 (1) — Skin (cellulitis)
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 1 (1)
Infection with unknown ANC - Bladder (urinary) (Infections and infestations) | 1 (1) — Bladder (urinary)
Leukocytes (total WBC) (Investigations) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Neurology - Other (Specify, __) (Nervous system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 3 (3)
Obstruction, GU - Bladder (Renal and urinary disorders) | 1 (1)
Pain - Abdomen NOS (Gastrointestinal disorders) | 2 (2)
Pain - Back (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Bladder (Renal and urinary disorders) | 1 (1)
Pain - Cardiac/heart (Cardiac disorders) | 1 (1)
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Chest/thorax NOS (General disorders) | 2 (2)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain - Head/headache (Nervous system disorders) | 2 (2)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Neck (Musculoskeletal and connective tissue disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 1 (2)
Platelets (Investigations) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Rigors/chills (General disorders) | 3 (4)
Supraventricular and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 3 (5)
Supraventricular and nodal arrhythmia - Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 2 (2)
Syndromes - Other (Specify, __) (General disorders) | 1 (1) — Systemic inflammatory response syndrome
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1)
Urine color change (Renal and urinary disorders) | 2 (2)
Vision-blurred vision (Eye disorders) | 1 (1)
Vision-flashing lights/floaters (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-azacytidine and Lintuzumab (N=7)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4 (11)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (7)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 2 (9)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 (3)
Anorexia (Gastrointestinal disorders) | 3 (7)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (7)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 2 (3)
Bilirubin (hyperbilirubinemia) (Investigations) | 3 (8)
Constipation (Gastrointestinal disorders) | 7 (29)
Constitutional Symptoms - Other (Specify, __) (General disorders) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (15)
Cytokine release syndrome/acute infusion reaction (Immune system disorders) | 1 (1)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 1 (4)
Diarrhea (Gastrointestinal disorders) | 4 (17)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7 (37)
Edema: head and neck (General disorders) | 1 (2)
Edema: limb (General disorders) | 4 (33)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 7 (52)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2 (4)
Flushing (Skin and subcutaneous tissue disorders) | 1 (2)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (5)
Hematoma (Vascular disorders) | 1 (4)
Hemoglobin (Blood and lymphatic system disorders) | 7 (41)
Hemorrhage, GI - Lower GI NOS (Gastrointestinal disorders) | 1 (3)
Hemorrhage/Bleeding - Other (Vascular disorders) | 1 (2)
Hot flashes/flushes (Vascular disorders) | 1 (6)
Hypotension (Vascular disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Incontinence, anal (Gastrointestinal disorders) | 1 (4)
Incontinence, urinary (Renal and urinary disorders) | 1 (2)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e (Infections and infestations) | 2 (7)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e (Infections and infestations) | 1 (3)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e (Infections and infestations) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 1 (1)
Infection with unknown ANC - Upper airway NOS (Infections and infestations) | 1 (2)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (25)
Leukocytes (total WBC) (Investigations) | 7 (31)
Lymphopenia (Investigations) | 4 (23)
Mood alteration - Anxiety (Psychiatric disorders) | 2 (20)
Mood alteration - Depression (Psychiatric disorders) | 2 (13)
Muscle weakness, generalized or specific area (not due to neuropathy) - Facial (Musculoskeletal and connective tissue disorders) | 1 (5)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 2 (9)
Nausea (Gastrointestinal disorders) | 5 (33)
Neurology - Other (Specify, __) (Nervous system disorders) | 1 (2)
Neuropathy: sensory (Nervous system disorders) | 1 (5)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 7 (33)
Ocular/Visual - Other (Specify, __) (Eye disorders) | 1 (1)
Pain - Abdomen NOS (Gastrointestinal disorders) | 2 (4)
Pain - Back (Musculoskeletal and connective tissue disorders) | 3 (15)
Pain - Cardiac/heart (Cardiac disorders) | 1 (2)
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1 (3)
Pain - Chest/thorax NOS (General disorders) | 1 (2)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 4 (17)
Pain - Eye (Eye disorders) | 1 (5)
Pain - Head/headache (Nervous system disorders) | 4 (22)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 3 (16)
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 2 (14)
Pain - Neck (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain - Other (Specify, __) (General disorders) | 4 (23)
Pain - Pain NOS (General disorders) | 2 (10)
Pain - Rectum (Gastrointestinal disorders) | 1 (9)
Pain - Sinus (Nervous system disorders) | 1 (2)
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Palpitations (Cardiac disorders) | 2 (5)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (7)
Platelets (Investigations) | 7 (48)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (6)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (3)
PTT (Partial Thromboplastin Time) (Investigations) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (13)
Rigors/chills (General disorders) | 4 (14)
Salivary gland changes/saliva (Gastrointestinal disorders) | 1 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 4 (12)
Supraventricular and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 3 (7)
Supraventricular and nodal arrhythmia - Supraventricular tachycardia (Cardiac disorders) | 1 (2)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 3 (14)
Syncope (fainting) (Nervous system disorders) | 1 (4)
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 1 (3)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1)
Urine color change (Renal and urinary disorders) | 2 (6)
Vision-blurred vision (Eye disorders) | 1 (3)
Vomiting (Gastrointestinal disorders) | 3 (10)
Watery eye (epiphora, tearing) (Eye disorders) | 1 (2)
Keratitis (corneal inflammation/corneal ulceration) (Eye disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was terminated early by the sponsor due to the removal of lintuzumab from the market.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No